CLINICAL TRIAL: NCT06306248
Title: Adjusting Immune Activation to Reinstate Neural Plasticity and Promote the Beneficial Effect of Non-pharmacological Interventions
Brief Title: Immune Activation, Neural Plasticity and Depression
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Sara Poletti, Principal Investigator, IRCCS Ospedale San Raffaele
Other Study IDs: PNRR-MAD-2022-12375716
Record Dates: First submitted 2024-02-27; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Mood Disorders; Major Depressive Disorder; Sleep Deprivation
MeSH Terms: conditions — Mood Disorders; Depressive Disorder, Major; Sleep Deprivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MDD patients: 60 patients with a depressive episode in course of major depression (MDD) and treated with a chronobiological intervention including total sleep deprivation (TSD) + light therapy (LT).
  Each subject will participate in the study for 6 months, will undergo MRI and clinical evaluation that will take overall about 2 hours at baseline (V0), after one week of chronobiological treatment and at 6 month follow-up.
  Interventions: Other: Total sleep deprivation

INTERVENTIONS:
Other: Total sleep deprivation — non pharmacologic treatment for depression

SUMMARY:
Major depressive disorder (MDD) is a chronic, recurring and potentially life-threatening illness that affects up to 10% of the population across the globe.Increasing evidence indicates a clear link between immune dysfunction and MDD.Moreover, an activation of inflammatory pathways is associated to a lack of clinical response to antidepressants. Thus, the regulation of inflammation represents a potential approach to modulate the link between the living environment and antidepressant outcome. Light therapy combined with sleep deprivation hastens recovery, with benefits that can be perceived by patients during the first week of treatment. Alteration of the sleep-wake cycle and of sleep structure are core symptoms of MDD.The aims of the present project are (i) to show that neural plasticity and the environmental context are moderating factors of the therapeutic outcome of immune modulation and (ii) to exploit their interplay to set up novel and effective therapeutic strategies for MDD.This is a observational prospective study with non-invasive add-on procedures (Magnetic Resonance without contrast). In this study, 60 patients with a depressive episode in course of MDD and treated with a chronobiological intervention including total sleep deprivation (TSD) + light therapy (LT), as performed in clinical practice, will be studied. All participants enrolled in the study will receive Treatment As Usual (TAU), i.e., pharmacotherapy, chronobiological intervention plus clinical management. Drug prescription will be performed during the clinical management sessions.The study will have a total duration of 24 months. Each subject will participate in the study for 6 months, will undergo Magnetic Resonance Imaging (MRI) and clinical evaluation at baseline, after one week of chronobiological treatment and at 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* A depressive episode according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria in the course of MDD with:

  * HDRS score > 17
  * Age 18-65 years;
  * In treatment with TSD+LT
* Signed informed consent, able to understand, speak and write the national language

Exclusion Criteria:

* History of bipolar disorder, schizophrenia, schizoaffective disorder, psychosis not otherwise specified; anorexia or bulimia nervosa;
* Taking following medications: antipsychotics, anticonvulsants, mood stabilizers; stimulants
* Active infection requiring antibiotics therapy;
* Immunosuppressed patient or other chronic diseases
* Signs of active infection requiring treatment
* Use of anti-inflammatory medication on a regular basis for a chronic inflammatory/autoimmune Disorder. Forbidden treatment: corticosteroids, Non Steroidal Anti-inflammatory Drugs, immunosuppressant IV-Ig based treatment
* Ongoing fever, infection treated by antibiotics or uncontrolled diabetes type I or II;
* Existing cancer or history of cancer in the last 5 years (except skin epidermoid cancer or in-situ cervix cancer);
* Known HIV infection or clinically manifest Acquired Immune Deficiency Syndrome (AIDS), Parkinson's or Alzheimer's disease, or any other serious condition likely to interfere e with the conduct of the trial;
* Abuse of drugs or alcohol in the past 6 months Other exclusion criteria related to the MRI procedure include
* Aneurysm clip
* Implanted neural stimulator
* Implanted cardiac pacemaker or auto-defibrillator
* Cochlear implant
* Ocular foreign body (e.g., metal shavings)
* Any implanted device (pumps, infusion devices, etc)
* Shrapnel injuries

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with major depressive disorder
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2025-03-03 (Estimated); Study Completion 2025-05-09 (Estimated)

PRIMARY OUTCOMES:
BENEFICIAL EFFECT OF total sleep deprivation in inflamed vs non inflamed patients. | at baseline, 1 week follow-up, 6 months follow up
  Response to total sleep deprivation will be measured (50% reduction in hamilton depression rating scale (HDRS), min score 0 max 52; higher scores higher severity of depression) in patients with C reactive protein levels <3 and >=3 mg/L.

SECONDARY OUTCOMES:
Neurobiological markers of prediction and progression of antidepressant treatment | from baseline to 6 months follow up
  a machine learning algorithm will be implemented to identify markers of prediction of response to treatment (50% reduction in HDRS, min score 0 max 52; higher scores higher severity of depression) and disease progression (number of relapses and severity of depression at 6 months follow-up) based on changes in peripheral inflammatory markers and in brain measures of neural plasticity (e.g. brain levels of glutamate and GABA; measures of resting state functional connectivity: amplitude of low-frequency fluctuation, regional homogeneity) and structural integrity (e.g. brain volumes, white matter microstructure - fractional anisotropy).

CONTACTS AND LOCATIONS:
Overall Officials: Sara Poletti, PhD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Mi, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trivedi MH, Rush AJ, Wisniewski SR, Nierenberg AA, Warden D, Ritz L, Norquist G, Howland RH, Lebowitz B, McGrath PJ, Shores-Wilson K, Biggs MM, Balasubramani GK, Fava M; STAR*D Study Team. Evaluation of outcomes with citalopram for depression using measurement-based care in STAR*D: implications for clinical practice. Am J Psychiatry. 2006 Jan;163(1):28-40. doi: 10.1176/appi.ajp.163.1.28. PMID 16390886
- [Background] Benedetti F, Dallaspezia S, Melloni EMT, Lorenzi C, Zanardi R, Barbini B, Colombo C. Effective Antidepressant Chronotherapeutics (Sleep Deprivation and Light Therapy) Normalize the IL-1beta:IL-1ra Ratio in Bipolar Depression. Front Physiol. 2021 Sep 1;12:740686. doi: 10.3389/fphys.2021.740686. eCollection 2021. PMID 34539454
- [Background] Miller AH, Raison CL. The role of inflammation in depression: from evolutionary imperative to modern treatment target. Nat Rev Immunol. 2016 Jan;16(1):22-34. doi: 10.1038/nri.2015.5. PMID 26711676
- [Background] Leboyer M, Berk M, Yolken RH, Tamouza R, Kupfer D, Groc L. Immuno-psychiatry: an agenda for clinical practice and innovative research. BMC Med. 2016 Oct 28;14(1):173. doi: 10.1186/s12916-016-0712-5. PMID 27788673
- [Background] Harrison NA, Brydon L, Walker C, Gray MA, Steptoe A, Critchley HD. Inflammation causes mood changes through alterations in subgenual cingulate activity and mesolimbic connectivity. Biol Psychiatry. 2009 Sep 1;66(5):407-14. doi: 10.1016/j.biopsych.2009.03.015. Epub 2009 May 7. PMID 19423079
- [Background] Hepgul N, Cattaneo A, Agarwal K, Baraldi S, Borsini A, Bufalino C, Forton DM, Mondelli V, Nikkheslat N, Lopizzo N, Riva MA, Russell A, Hotopf M, Pariante CM. Transcriptomics in Interferon-alpha-Treated Patients Identifies Inflammation-, Neuroplasticity- and Oxidative Stress-Related Signatures as Predictors and Correlates of Depression. Neuropsychopharmacology. 2016 Sep;41(10):2502-11. doi: 10.1038/npp.2016.50. Epub 2016 Apr 12. PMID 27067128
- [Background] Carvalho LA, Torre JP, Papadopoulos AS, Poon L, Juruena MF, Markopoulou K, Cleare AJ, Pariante CM. Lack of clinical therapeutic benefit of antidepressants is associated overall activation of the inflammatory system. J Affect Disord. 2013 May 15;148(1):136-40. doi: 10.1016/j.jad.2012.10.036. Epub 2012 Nov 27. PMID 23200297
- [Background] Branchi I, Poggini S, Capuron L, Benedetti F, Poletti S, Tamouza R, Drexhage HA, Penninx BWJH, Pariante CM; European College of Neuropsychopharmacology (ECNP) ImmunoNeuroPsychiatry Thematic Working Group and Marion Leboyer. Brain-immune crosstalk in the treatment of major depressive disorder. Eur Neuropsychopharmacol. 2021 Apr;45:89-107. doi: 10.1016/j.euroneuro.2020.11.016. Epub 2020 Dec 29. PMID 33386229
- [Background] Dinan TG. Inflammatory markers in depression. Curr Opin Psychiatry. 2009 Jan;22(1):32-6. doi: 10.1097/YCO.0b013e328315a561. PMID 19122532
- [Background] Otte C, Gold SM, Penninx BW, Pariante CM, Etkin A, Fava M, Mohr DC, Schatzberg AF. Major depressive disorder. Nat Rev Dis Primers. 2016 Sep 15;2:16065. doi: 10.1038/nrdp.2016.65. PMID 27629598
- [Background] Kohler O, Benros ME, Nordentoft M, Farkouh ME, Iyengar RL, Mors O, Krogh J. Effect of anti-inflammatory treatment on depression, depressive symptoms, and adverse effects: a systematic review and meta-analysis of randomized clinical trials. JAMA Psychiatry. 2014 Dec 1;71(12):1381-91. doi: 10.1001/jamapsychiatry.2014.1611. PMID 25322082
- [Background] Muller N, Schwarz MJ, Dehning S, Douhe A, Cerovecki A, Goldstein-Muller B, Spellmann I, Hetzel G, Maino K, Kleindienst N, Moller HJ, Arolt V, Riedel M. The cyclooxygenase-2 inhibitor celecoxib has therapeutic effects in major depression: results of a double-blind, randomized, placebo controlled, add-on pilot study to reboxetine. Mol Psychiatry. 2006 Jul;11(7):680-4. doi: 10.1038/sj.mp.4001805. Epub 2006 Feb 21. PMID 16491133
- [Background] Wittenberg GM, Stylianou A, Zhang Y, Sun Y, Gupta A, Jagannatha PS, Wang D, Hsu B, Curran ME, Khan S; MRC ImmunoPsychiatry Consortium; Chen G, Bullmore ET, Drevets WC. Effects of immunomodulatory drugs on depressive symptoms: A mega-analysis of randomized, placebo-controlled clinical trials in inflammatory disorders. Mol Psychiatry. 2020 Jun;25(6):1275-1285. doi: 10.1038/s41380-019-0471-8. Epub 2019 Aug 19. PMID 31427751
- [Background] Warner-Schmidt JL, Vanover KE, Chen EY, Marshall JJ, Greengard P. Antidepressant effects of selective serotonin reuptake inhibitors (SSRIs) are attenuated by antiinflammatory drugs in mice and humans. Proc Natl Acad Sci U S A. 2011 May 31;108(22):9262-7. doi: 10.1073/pnas.1104836108. Epub 2011 Apr 25. PMID 21518864
- [Background] Dallaspezia S, Benedetti F. Chronobiological therapy for mood disorders. Expert Rev Neurother. 2011 Jul;11(7):961-70. doi: 10.1586/ern.11.61. PMID 21721914
- [Background] WHO, 2008 The global burden of disease: 2004 update